CLINICAL TRIAL: NCT05866861
Title: A Phase Ib, Randomized, Double-Blind, Placebo-Controlled, Ascending-Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Subcutaneously Administered CUG252 Following Multiple Dose Administrations in Participants With Mild-to-Moderate SLE
Brief Title: A Study in Participants With Mild-to-moderate Systemic Lupus Erythematosus
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Cugene Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CUG252-P102
Record Dates: First submitted 2023-03-20; First posted 2023-05-19 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Systemic Lupus Erythematosus; SLE (Systemic Lupus); Autoimmune
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- CUG252 (Experimental): CUG252 or placebo will be administered to participants in a 3:1 ratio.
  Interventions: Drug: CUG252
- Placebo (Placebo Comparator): CUG252 or placebo will be administered to participants in a 3:1 ratio.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CUG252 — CUG252 will be administered by subcutaneous injection.
  Arms: CUG252
Drug: Placebo — Placebo will be administered by subcutaneous injection.
  Arms: Placebo

SUMMARY:
The main purpose of this study is to evaluate the safety and tolerability of CUG252 following multiple ascending doses in participants with Systemic Lupus Erythematosus (SLE).

DETAILED DESCRIPTION:
CUG252 is a potential best-in-class engineered IL-2 compound, designed to have improved Treg selectivity while reducing undesired IL-2 activity.

This study will evaluate safety, tolerability, pharmacokinetics (PK), pharmacodynamics (PD), and immunologic effects of CUG252 following subcutaneous administration of multiple ascending doses in participants with mild-to-moderate SLE. The effects of SLE disease activity and biomarkers will also be evaluated.. The SLE participants will receive randomized multiple subcutaneous doses of CUG252 or placebo. After receiving the last dose of CUG252 or placebo, participants will be followed to study day 64 post first dose administration to evaluate safety, PK, PD and preliminary efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Male or female participant, aged 18 to 65 years (inclusive), at time of consent
* BMI greater than or equal to 18 and less than 39 kg/m2 at Screening
* Diagnosis of SLE at least 6 months prior to Screening
* Minimal to moderate SLE disease activity
* If a participant is taking oral prednisone, the dose must be less than or equal to 20 mg/day for a minimum of 8 weeks prior to Screening and at a stable dose for a minimum of 2 weeks prior to Screening
* If a participant is taking azathioprine, antimalarial, mycophenolate mofetil, or methotrexate, the medication(s) must have been started a minimum of 12 weeks prior to Screening and at a stable dose for a minimum of 8 weeks prior to Screening

Exclusion Criteria:

* Have one or more of the following medical conditions: SARS-CoV-2 infection 30 days prior to drug administration, evidence of Grade 3 or greater hematologic, hepatic, or rental dysfunction, active severe or unstable neuropsychiatric SLE, active severe renal disease, history of severe active lupus nephritis with proteinuria levels greater than 1.0 g/24 hours, or dialysis in the last 6 months. History of current diagnosis of other autoimmune/inflammatory diseases, history of any non-SLE disease that has required treatment with corticosteroids for more than 2 weeks within the last 12 weeks prior to Screening, active clinically significant bacterial, viral, or fungal infection at Screening, active or latent TB at Screening, pulmonary infection or active lung disease besides those related to lupus, or severe pulmonary disease requiring oxygen therapy. History of condition that predisposes participant to infection, confirmed positive serology at Screening, history of opportunistic infection requiring hospitalization or IV antimicrobial treatment within the last year, history of organ or hematopoietic stem cell transplant, history of major surgery within 12 weeks of Screening, history of significant cardiovascular disease, history of gastrointestinal bleeding, history of cancer apart from successfully treated squamous or basal cell carcinoma or cervical cancer in situ.
* Are on one or more of the following medications: have received vaccination within 30 days prior to Screening (including COVID-19 vaccination), Aldesleukin or other IL-2 derivatives at any time, T cell depleting agents and inhibitors of T cell activation at any time, Anti-BLyS/BAFF inhibitors, IL-1 receptor antagonist, anti-TNF therapy, and anti-interferon alpha receptor inhibitor within 3 months prior to Screening, rituximab or other B-cell depleting agent within 6 months, glucocorticoids within 6 weeks prior to Day 1, other immunosuppressant drugs within 8 weeks, history of cytotoxic medications within 12 months, receipt of blood products within 6 months, plasmapheresis within 30 days of Screening.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2023-04-24 (Actual); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
Number and percentage of subjects with Treatment Emergent Adverse Events | Up to 64 Days
  To evaluate the safety and tolerability of multiple ascending doses (MAD) in participants with mild to moderate SLE.

SECONDARY OUTCOMES:
Pharmacokinetics profile of CUG252 (AUC) | Day 1 pre dose through Day 64
  To assess the Area under the plasma concentration versus time curve (AUC)
Pharmacokinetics profile of CUG252 (Cmax) | Day 1 pre dose through Day 64
  To assess the maximum plasma concentration (Cmax)
Pharmacokinetics profile of CUG252 (Tmax) | Day 1 pre dose through Day 64
  To assess the time of maximum concentration (Tmax)
Pharmacokinetics profile of CUG252 (t1/2) | Day 1 pre dose through Day 64
  To assess the half-life (t1/2)
Immunogenicity of CUG252 | Day 1 pre dose through Day 64
  To measure the serum concentration of antibodies against CUG252
Change in the number and percentages of immune cells | Day 1 pre dose through Day 64
  To assess the effect of CUG252 on immuno-pharmacodynamic endpoints.

CONTACTS AND LOCATIONS:
Locations (11):
- United States (11):
  - Site 1001, Anniston, Alabama
  - Site 1011, La Jolla, California
  - Site 1002, Clearwater, Florida
  - Site 1009, Tampa, Florida
  - Site 1007, Lawrenceville, Georgia
  - Site 1010, Columbus, Ohio
  - Site 1005, Middleburg Heights, Ohio
  - Site 1003, Duncansville, Pennsylvania
  - Site 1006, Dallas, Texas
  - Site 1004, Mesquite, Texas
  - Site 1012, Seattle, Washington